CLINICAL TRIAL: NCT01930123
Title: Impact of Fructose on Metabolism, Energy Homeostasis and Magnetic Resonance (MR) Biomarkers in Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Impact of Fructose on Metabolism, Energy Homeostasis and Magnetic Resonance Biomarkers in Nonalcoholic Fatty Liver Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: Manal F Abdelmalek (Other)
Responsible Party: Sponsor-Investigator, Manal F Abdelmalek, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00031687
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: Fructose; NASH; advanced fibrosis; biomarker; magnetic resonance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with NAFLD (Experimental): 70 subjects with biopsy-proven NAFLD; subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  Interventions: Drug: intravenous fructose challenge; Other: Blood Draw
- Health controls (Active Comparator): 15 healthy controls for comparison with NAFLD patients.The 15 subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  Interventions: Drug: intravenous fructose challenge; Other: Blood Draw

INTERVENTIONS:
Drug: intravenous fructose challenge — Patients will be admitted to our Duke Clinical Research Unit (DCRU) at least 12 hours prior to morning intravenous fructose challenge. All patients will have a "standard" meal in order to control for dietary composition and calorie intake prior to intravenous fructose challenge. Patients will be NPO (nothing by mouth) after midnight for morning IV fructose MR biomarker measures. Patients with suspected NAFLD will have had an historical standard of care liver biopsy in the past and will have IV fructose Magnetic Resonance biomarker measures in the morning.
Other: Blood Draw — Fasting bloodwork will be obtained before and after the IV fructose challenge.

SUMMARY:
This study will advance several goals of the NIH Action Plan: 1) establish a multidisciplinary team to develop quantitative methodologies and imaging protocols for liver, 2) validate diagnostic criteria and methodologies for imaging in liver in both a cross-sectional and a longitudinal dietary intervention study of patients with Nonalcoholic Fatty Liver Disease (NAFLD), 3) create a liver tissue bank with correlative imaging data, 4) develop reliable non-invasive MR markers to distinguish simple steatosis from Nonalcoholic Steatohepatitis (NASH), and 5) define the dynamic changes in metabolism, energy homeostasis, and MR biomarkers as they relate to fructose-related liver injury.

DETAILED DESCRIPTION:
Like obesity, NAFLD and NASH are closely linked to nutrition and the "Western diet" which is rich in saturated fats and refined sugars. Although fat consumption has remained relatively stable, the marked increase in dietary fructose consumption (more than doubling in the past 30 years alone) supports the role of fructose in NAFLD and the metabolic syndrome. Although the mechanism(s) for fructose-related liver injury is not yet well defined, fructose-related hepatic adenosine triphosphate (ATP) depletion may contribute to liver injury. Observations in animals suggest that fructose induces metabolic syndrome and NAFLD independent of energy intake. One key difference in fructose metabolism (as opposed to glucose) relates to ATP depletion and the necessity of adenosine monophosphate (AMP) kinase to replenish ATP stores. As opposed to glucose, initial fructose metabolism involves phosphorylation of fructose to fructose-1-phosphate by fructokinase (ketohexokinase, KHK) using the substrate ATP. Unlike glucokinase, the phosphorylation of fructose by KHK is specific for fructose and not rate limited. Replenishment of ATP stores requires phosphorylation of AMP back to ATP via AMP kinase (which is inhibited in insulin resistance (common in patients with NAFLD) or conversion to uric acid via xanthine dehydrogenase resulting in hyperuricemia. The high activity of KHK in phosphorylating fructose to fructose-1-phosphate in the liver, could result in hepatic ATP depletion with habitual fructose consumption.

Published animal and human studies support our hypothesis that fructose is a risk factor for NAFLD and NAFLD-related liver disease progression. In animal models, diets high in fructose induce features of the metabolic syndrome including weight gain, insulin resistance, hypertriglyceridemia, and hypertension. Similar effects are not observed with the administration of other simple sugars such as glucose. Fructose (or sucrose) administration to humans also causes features of metabolic syndrome which are quite typical of patients with NAFLD. Fructose is lipogenic, stimulates triglyceride synthesis and causes hepatic steatosis. As previously reported in animals, our group reported that increased fructose consumption (assessed as fructose-containing beverages only) is a risk factor of metabolic syndrome and biopsy-proven NAFLD and that patients with NAFLD consume 3-4 times more fructose than age, gender, and mass index (BMI) matched controls without liver disease.

In addition to increased fructose consumption being a risk factor for NAFLD, fructose has been implicated in NAFLD disease progression. The administration of a diet with 25% of total energy as sucrose (which contains 50% fructose) resulted in a rise in liver aminotransferase levels within 18 days. This study, performed nearly 25 years ago, is all the more alarming as current sugar intake of Americans is in this same range. In our study of 427 patients with biopsy-proven NAFLD, increased consumption of fructose-containing beverages was univariately associated with decreased age (P < 0.0001), male sex (P < 0.0001), hypertriglyceridemia (P < 0.04), low high density lipoprotein (HDL) cholesterol (<0.0001), decreased serum glucose (P < 0.001), increased calorie intake (P < 0.0001), and hyperuricemia (P < 0.0001). After controlling for age, sex, BMI, and total calorie intake, daily fructose consumption was associated with lower steatosis grade and higher fibrosis stage (P < 0.05 for each). Being that triglyceride synthesis requires ATP, we hypothesize that lower hepatic steatosis may reflect deceased ATP availability. Additionally, in older adults (age ≥ 48 years), daily fructose consumption was associated with increased hepatic inflammation (P < 0.05), and hepatocyte ballooning (P< 0.05). However, the mechanism(s) by which fructose causes liver injury remains unknown.

In support of our hypothesis that ATP depletion underlies liver injury in patients with NAFLD, our group has demonstrated that patients with biopsy-proven NAFLD have increased hepatic mRNA (messenger ribonucleic acid) expression of KHK compared to matched controls. Indeed, in human pilot studies, intravenous (IV) fructose administration is associated with hepatic ATP depletion which can be assessed by 31P magnetic resonance spectroscopy (MRS). Reduced hepatic ATP stores are more prevalent in overweight and obese subjects than in lean subjects. Furthermore, recovery from fructose-induced ATP depletion was found to be delayed in patients with NAFLD (n=8). However, a limitation to this existing work is the small sample size and the inability to assess a cause-effect relationship(s) between BMI, NAFLD, energy homeostasis, and histologic features of liver injury. In liver cells, ATP depletion could perpetuate chronic liver injury by making fatty hepatocytes less proliferative. Hepatic ATP depletion also encourages the expansion of liver progenitor populations, causes arrest in protein synthesis, induces inflammatory and prooxidative changes, increases endoplasmic reticulum stress, promotes activation of stress-related kinases, induces mitochondrial dysfunction, and increases apoptotic activity. This supporting data suggests that fructose may be associated with NAFLD, NASH, and progressive fibrosis. Further, a study by Loguercio et al. demonstrated that increased uric acid levels above the basal level after IV fructose infusion was significantly higher (p < 0.01) in patients with cirrhosis (3 mg/dl) and NASH (1.9 mg/dl) than in healthy controls (1.2 mg/dl). This effect was completely reversed by fructose 1,6-diphosphate which could replenish the ability to resynthesize ATP (adenosine triphosphate) from ADP (adenosine diphosphate). Therefore, an IV fructose challenge could effectively differentiate healthy subjects, from chronic hepatitis, from cirrhosis.

NAFLD lacks accurate and robust non-invasive biomarkers to grade and stage histologic disease activity. This is a critical barrier to understanding the influence of this important environmental risk factor (increased/habitual fructose consumption) on the pathogenesis and progression of NAFLD. Currently, reliable assessment NAFLD requires liver biopsy and interpretation of histology. Serum aminotransferase levels and conventional imaging methods can detect liver fat but cannot grade or stage NAFLD. Furthermore, current developments in biomarker are cross-sectional in nature and do not characterize the dynamic changes which underlie liver injury in patients with NAFLD. In vivo 31P MRS permits the evaluation of dynamic changes of individual phosphorus-containing metabolites in the liver parenchyma, such as phosphomonoester (PME), ATP, and inorganic phosphate (Pi). Intravenous fructose load alters phosphorus metabolites and allows assessment of liver function by 31P MRS. Other investigators have demonstrated that fructose loading could be used effectively as a tool to investigate change in metabolic steps of hepatic metabolism in humans with alcohol-related liver disease. Further, IV fructose loading causes significantly higher ATP degradation and uric acid production in cirrhotic patients than in healthy controls. The associations between fructose, increased uric acid, and hepatic ATP depletion has been previously described. Increased uric acid is an independent risk factor for NAFLD and in keeping with our hypothesis, hyperuricemia may be a surrogate marker of impaired hepatic energy homeostasis in patients with NAFLD. The proposed mechanism for fructose-related hepatic ATP depletion, NAFLD, NASH and the associated hyperuricemia is depicted in Figure 1 is novel, innovative, scientifically rigorous and address an important public health concern-the impact of fructose on the rising epidemic of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following criteria to be eligible for enrollment:

* Age greater than 18 years as of the initial screening interview and provision of consent
* Healthy control as defined by:

  * normal liver aminotransferases AND
  * no evidence of NAFLD on radiologic imaging studies AND
  * no history of chronic liver disease OR
  * liver biopsy (if one had been historically performed for evaluation of suspected liver disease).

OR • Patient with clinically suspected NAFLD as assessed by standard of care measures (risk factors for NAFLD, abnormal liver enzymes and/or fatty liver on imaging studies) who are scheduled to will undergo liver biopsy for the purpose of grading / staging the severity of their underlying liver disease

Exclusion Criteria:

Patients who satisfy any of the following exclusion criteria will be ineligible for enrollment:

* Current or history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening (significant alcohol consumption is defined as more than 20 g/day in females and more than 30 g/day in males, on average)
* Inability to reliably quantify alcohol consumption based upon local study physician judgment
* Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the past year prior to randomization
* Prior or planned (during the study period) bariatric surgery
* Uncontrolled diabetes defined as HbA1c 9.5% or higher within 60 days prior to enrollment
* A platelet count below 90,000/mm3
* Clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities:

  * Serum albumin greater than 3.2 g/dL, INR (international normalized ratio) greater than 1.3, bilirubin greater than 2.0 mg/dL
  * History of esophageal varices, ascites or hepatic encephalopathy
* Evidence of other forms of chronic liver disease
* Serum alanine aminotransferase (ALT) greater than 300 U/L
* Serum creatinine of 2.0 mg/dL or greater
* Unstable therapy for components of the metabolic syndrome (ie. recent starting or stopping of insulin sensitizing agent, lipid lowering agent, and/or antioxidant therapy) . Recent starting or stopping (for more than 7 days) the use of a thiazolidinedione (pioglitazone or rosiglitazone) 90 days before the entry biopsy or anytime thereafter
* Use of any prescription or over-the-counter medication or herbal remedy that are believed to improve or treat NASH or liver disease or obesity for the 90 days prior to baseline liver biopsy or prior to randomization

  - Patients must not take any other agent to treat NASH except the treatment assigned after randomization.
* Inability to safely obtain a liver biopsy
* Active substance abuse including inhaled or injection drugs in the year prior to screening
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial, breast feeding
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* A contraindication to MRI examinations
* Extreme claustrophobia
* Weight or girth exceeds the scanner capabilities
* Any condition or circumstance that, in the opinion of the site investigator, would interfere with completion of MR examinations
* Failure to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-10; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manal F Abdelmalek, MD., MPH, Principal Investigator — DUMC - Gastroenterology; Brian Soher, PhD, Principal Investigator — DUMC -Radiology; Mustafa Bashir, MD, Principal Investigator — DUMC - Radiology; Cynthia Guy, MD, Principal Investigator — DUMC- Pathology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited prior to liver biopsy between November 2014 and January 2020.
Groups:
- Patients With NAFLD: Subjects with biopsy-proven NAFLD; subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  intravenous fructose challenge: Patients will be admitted to our Duke Clinical Research Unit (DCRU) at least 12 hours prior to morning intravenous fructose challenge. All patients will have a "standard" meal in order to control for dietary composition and calorie intake prior to intravenous fructose challenge. Patients will be NPO (nothing by mouth) after midnight for morning IV fructose MR biomarker measures. Patients with suspected NAFLD will have had an historical standard of care liver biopsy in the past and will have IV fructose Magnetic Resonance biomarker measures in the morning.
  Blood Draw: Fasting bloodwork will be obtained before and after the IV fructose challenge.
- Healthy Controls: Healthy controls for comparison with NAFLD patients.The 15 subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  Intravenous fructose challenge: Patients will be admitted to our Duke Clinical Research Unit (DCRU) at least 12 hours prior to morning intravenous fructose challenge. All patients will have a "standard" meal in order to control for dietary composition and calorie intake prior to intravenous fructose challenge. Patients will be NPO (nothing by mouth) after midnight for morning IV fructose MR biomarker measures. Patients with suspected NAFLD will have had an historical standard of care liver biopsy in the past and will have IV fructose Magnetic Resonance biomarker measures in the morning.
  Blood Draw: Fasting bloodwork will be obtained before and after the IV fructose challenge.
Period: Overall Study
Arm/Group | Patients With NAFLD | Healthy Controls
Started | 81 | 37
Completed | 58 | 29
Not Completed | 23 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 21 | 8
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Groups:
- Healthy Controls: 15 healthy controls for comparison with NAFLD patients.The 15 subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  intravenous fructose challenge: Patients will be admitted to our Duke Clinical Research Unit (DCRU) at least 12 hours prior to morning intravenous fructose challenge. All patients will have a "standard" meal in order to control for dietary composition and calorie intake prior to intravenous fructose challenge. Patients will be NPO (nothing by mouth) after midnight for morning IV fructose MR biomarker measures. Patients with suspected NAFLD will have had an historical standard of care liver biopsy in the past and will have IV fructose Magnetic Resonance biomarker measures in the morning.
  Blood Draw: Fasting bloodwork will be obtained before and after the IV fructose challenge.
- Total: Total of all reporting groups
Arm/Group | Patients With NAFLD | Healthy Controls | Total
Number analyzed (Participants) | 58 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (10.2) | 38.0 (16.9) | 48.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 16 | 55
  Male | 19 | 13 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 56 | 28 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 47 | 22 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 29 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Glucose Level From Pre-fructose Administration to Post-fructose Administration in Control Cohort
Time Frame: Baseline to approximately one hour post-fructose administration
Population: Not applicable to the Patients with NAFLD arm. Data collected on 19 healthy controls.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Healthy Controls: Healthy controls for comparison with NAFLD patients. The subjects will be challenged with a fructose infusion after a period for 12 hours fasting.
  intravenous fructose challenge: Patients will be admitted to our Duke Clinical Research Unit (DCRU) at least 12 hours prior to morning intravenous fructose challenge. All patients will have a "standard" meal in order to control for dietary composition and calorie intake prior to intravenous fructose challenge. Patients will be NPO (nothing by mouth) after midnight for morning IV fructose MR biomarker measures. Patients with suspected NAFLD will have had an historical standard of care liver biopsy in the past and will have IV fructose Magnetic Resonance biomarker measures in the morning.
  Blood Draw: Fasting bloodwork will be obtained before and after the IV fructose challenge.
Arm/Group | Patients With NAFLD | Healthy Controls
Number analyzed (Participants) | 0 | 19
mg/dL |  | 6.26 (9.98)
Statistical Analysis 1: Comparison: Healthy Controls; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 6.26, Standard Deviation 9.98

2. Primary Outcome: Fructose-induced Change in Low Density Lipoproteins (LDL) Level
Description: Comparison between participants with mild fibrosis and participants with advanced fibrosis per the NAFLD Fibrosis score. The NAFLD Fibrosis score is a non-invasive scoring system based on several laboratory tests that helps to estimate the amount of scarring in the liver. A score of F0 or F1 is considered mild, F2 is indeterminate, and F3 or F4 is considered advanced.
Time Frame: Baseline to approximately one hour post-fructose administration
Population: Participants with mild or advanced fibrosis. Not applicable to the healthy controls arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Patients With NAFLD | Healthy Controls
Number analyzed (Participants) | 33 | 0
mg/dL
  NAFLD mild fibrosis: number analyzed (Participants) | 17 | 0
  NAFLD mild fibrosis | 5.47 (6.4) |
  NAFLD advanced fibrosis: number analyzed (Participants) | 16 | 0
  NAFLD advanced fibrosis | -1.13 (6.85) |
Statistical Analysis 1: Comparison: Patients With NAFLD; Mild fibrosis vs. advanced fibrosis; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Dynamic 31P Changes in Liver Beta-ATP Due to Fructose Injection
Description: Percent change of beta-ATP from baseline levels to lowest level (nadir) were evaluated in both controls and NAFLD subjects. 31P-MRS (magnetic resonance spectroscopy) measurements made every 90 seconds.
Time Frame: 6 Baseline measurements (~3 min), fructose injection and then approximately 30-50 minutes of 31P MRS with scans at 90 seconds
Population: Participants who had sufficient quality of MRS data.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Patients With NAFLD | Healthy Controls
Number analyzed (Participants) | 30 | 10
percentage of change | 56.7 (2.6) | 47.9 (5.2)
Statistical Analysis 1: Comparison: Patients With NAFLD vs Healthy Controls; Test type: Other; p = 0.09, t-test, 1 sided; Median Difference (Final Values) = 56.7, Standard Deviation 2.6

ADVERSE EVENTS:
Time Frame: up to 24 hours
Arm/Group | Patients With NAFLD | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/37
Other Adverse Events (participants affected / at risk) | 1/81 | 0/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With NAFLD (N=81) | Healthy Controls (N=37)
Swelling (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT01930123/Prot_SAP_000.pdf